CLINICAL TRIAL: NCT00150176
Title: A Randomized, Placebo-Controlled, Double-Blind Trial of Asenapine in the Prevention of Relapse After Long-Term Treatment of Schizophrenia
Brief Title: To Determine Long Term Efficacy and Safety of Asenapine in Schizophrenic Patient Population (A7501012)(COMPLETED)(P05770)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05770; A7501012
Record Dates: First submitted 2005-09-02; First posted 2005-09-08 (Estimated); Results first posted 2010-05-28 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asenapine (Experimental)
  Interventions: Drug: Asenapine - Open Label; Drug: Asenapine - Double Blind
- placebo (Placebo Comparator)
  Interventions: Drug: Asenapine - Open Label; Drug: Placebo - Double Blind

INTERVENTIONS:
Drug: Asenapine - Open Label — Open Label Phase: All subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1).
  Other Names: Saphris, Org 5222, SCH 900274
Drug: Placebo - Double Blind — Double Blind Phase: Following Open Label Phase, matching placebo sublingual twice daily for 26 weeks.
  Arms: placebo
Drug: Asenapine - Double Blind — Double Blind Phase: Following the Open Label Phase, asenapine 5 or 10 mg sublingual twice daily for 26 weeks.
  Other Names: Org 5222, SCH 900274, Saphris
  Arms: asenapine

SUMMARY:
Schizophrenia is a brain disease. The condition may be associated with acute psychotic episodes and long-term disability despite remission from the acute symptoms. Current management of schizophrenia focuses on the treatment of acute symptoms as well as long-term treatment aimed at preventing relapse after patients have experienced an improvement in acute symptoms. Patients who discontinue treatment have a high likelihood of experiencing relapse within 1-2 years after an acute episode of schizophrenia. Patients who remain on antipsychotic treatment have lower rates of relapse and have milder courses of exacerbation when relapse occurs.The symptoms of schizophrenia may be due to an imbalance in chemicals in the brain, primarily dopamine and serotonin, which enables brain cells to communicate with each other. Asenapine may help to correct the imbalance in dopamine and serotonin. The purpose of this clinical trial is to evaluate the efficacy of asenapine in preventing relapse/impending relapse (hereafter referred to as 'relapse') in subjects who have been treated with asenapine for symptoms of schizophrenia for 26 weeks. In addition, to determine the safety and tolerability of asenapine for up to 1-year of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a primary diagnosis of schizophrenia
* History of at least 1 prior episode of acute schizophrenia in the 3 years preceding screening
* History of schizophrenia requiring continuous antipsychotic treatment for at least 1 years preceding screening
* Clinically stable at the time of entry defined by at least a 4 week period of stable symptoms

Key Exclusion Criteria:

* Have an uncontrolled, unstable clinically significant medical condition
* History of suicide attempt or significant violence to others in the past 2 years
* A substance-induced psychotic disorder or behavioral disturbance thought to be due to substance abuse
* Current substance abuse/dependence
* Concurrent psychiatric disorder other than schizophrenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2005-04; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

REFERENCES:
- [Derived] Kane JM, Mackle M, Snow-Adami L, Zhao J, Szegedi A, Panagides J. A randomized placebo-controlled trial of asenapine for the prevention of relapse of schizophrenia after long-term treatment. J Clin Psychiatry. 2011 Mar;72(3):349-55. doi: 10.4088/JCP.10m06306. Epub 2011 Feb 22. PMID 21367356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, there was a 26 week open-label phase where 700 subjects received at least one dose of open-label asenapine (out of 831 initially enrolled). Only subjects who had continued stable presentation of symptoms during this phase were randomized into the double-blind phase.
Groups:
- Asenapine: Double Blind Asenapine Group. Subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1), followed by asenapine 5 or 10 mg sublingual twice daily for 26 weeks in the double blind phase.
- Placebo: Double Blind Placebo Group. Subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1), followed by matching placebo sublingual twice daily for 26 weeks during the double-blind phase.
Period: Overall Study
Arm/Group | Asenapine | Placebo
Started | 194 (subjects who were screened and received at least one dose of double-blind trial medication) | 192 (subjects who were screened and received at least one dose of double-blind trial medication)
Completed | 135 | 72
Not Completed | 59 | 120
Not completed — Adverse Event | 16 | 53
Not completed — Relapse/Impending relapse, non-AE | 10 | 39
Not completed — Withdrawal by Subject | 19 | 12
Not completed — Lost to Follow-up | 3 | 3
Not completed — OTHER | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Asenapine: Baseline for the double-blind period. Subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1), followed by asenapine 5 or 10 mg sublingual twice daily for 26 weeks in the double blind phase.
- Placebo: Baseline for the double-blind period. Subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1), followed by matching placebo sublingual twice daily for 26 weeks during the double-blind phase.
- Total: Total of all reporting groups
Arm/Group | Asenapine | Placebo | Total
Number analyzed (Participants) | 194 | 192 | 386
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (12.53) | 38.7 (11.64) | 38.9 (12.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 76 | 165
  Male | 105 | 116 | 221

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse or an Impending Relapse
Description: A relapse or impending relapse was declared if a subject meets 1 of 3 "symptomatic relapse criteria" which were all based on a combination of the Positive and Negative Syndrome Scale (PANSS) total score or PANSS items, and Clinical Global Impression-Severity (CGI-S); or if in the opinion of the investigator, the subject's symptoms of schizophrenia had deteriorated to such an extent or the risk of violence to self or others or risk of suicide had increased so that certain prespecified measures were necessary.
Time Frame: time of first relapse up to Day 182 (double blind phase)
Population: ITT population, excluding subjects not treated and w/ past enrollment in an asenapine trial. As trial progressed & subjects discont'd for various reasons, subjects at risk for relapse decreased from 190 each arm (Day 1) to 70 at risk in placebo arm and 135 subjects in asenapine arm (Day 182). Those relapsing >3 days after last dose also excluded.
Measure: Number; unit: relapses
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 190 | 190
relapses
  Days 1 - 7 (N asenapine = 190; N placebo = 190) | 0 | 3
  Days 8 - 14 (N asenapine = 188; N placebo = 186) | 1 | 14
  Days 15 - 21 (N asenapine = 183; N placebo = 170) | 2 | 9
  Days 22 - 28 (N asenapine = 180; N placebo = 160) | 2 | 8
  Days 29 - 35 (N asenapine = 175; N placebo = 149) | 0 | 7
  Days 36 - 42 (N asenapine = 175; N placebo = 140) | 1 | 8
  Days 43 - 49 (N asenapine = 173; N placebo = 130) | 5 | 2
  Days 50 - 56 (N asenapine = 166; N placebo = 127) | 1 | 4
  Days 57 - 63 (N asenapine = 165; N placebo = 123) | 1 | 1
  Days 64 - 70 (N asenapine = 163; N placebo = 120) | 2 | 3
  Days 71 - 77 (N asenapine = 161; N placebo = 117) | 1 | 4
  Days 78 - 84 (N asenapine = 160; N placebo = 113) | 2 | 2
  Days 85 - 91 (N asenapine = 158; N placebo = 110) | 0 | 4
  Days 92 - 98 (N asenapine = 154; N placebo = 104) | 0 | 4
  Days 99 - 105 (N asenapine = 151; N placebo = 99) | 0 | 2
  Days 106 - 112 (N asenapine = 151; N placebo = 96) | 0 | 1
  Days 113 - 119 (N asenapine = 149; N placebo = 95) | 2 | 3
  Days 120 - 126 (N asenapine = 147; N placebo = 87) | 0 | 1
  Days 127 - 133 (N asenapine = 147; N placebo = 86) | 0 | 1
  Days 134 - 140 (N asenapine = 146; N placebo = 84) | 0 | 0
  Days 141 - 147 (N asenapine = 145; N placebo = 83) | 0 | 1
  Days 148 - 154 (N asenapine = 142; N placebo = 81) | 0 | 5
  Days 155 - 161 (N asenapine = 141; N placebo = 75) | 0 | 1
  Days 162 - 168 (N asenapine = 139; N placebo = 74) | 1 | 0
  Days 169 - 175 (N asenapine = 137; N placebo = 72) | 2 | 1
  Days 176 - 182 (N asenapine = 135; N placebo = 70) | 0 | 1
  Days 183 - 189 (N asenapine = 75; N placebo = 39) | 0 | 0
  Days 190 - 196 (N asenapine = 9; N placebo = 9) | 0 | 0
  Days 197 - 203 (N asenapine = 2; N placebo = 2) | 0 | 0
  Days 204 - 210 (N asenapine = 0; N placebo = 1) | 0 | 0

2. Secondary Outcome: Time to Early Discontinuation for Any Reason
Description: The number of days to early discontinuation is the number of days from randomization to early discontinuation from the study for adverse event, relapse or impending relapse that was not considered an adverse event, withdrawal of informed consent, or lost to follow-up (without evidence of relapse).
Time Frame: time of discontinuation up to Day 182 (double blind phase)
Population: Intent to treat (ITT) population, additionally excluding subjects not treated and excluding subjects with past enrollment in an asenapine trial.
Measure: Number; unit: participants
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 191 | 191
participants
  Days 1 - 7 (N asenapine = 191; N placebo = 191) | 1 | 2
  Days 8 - 14 (N asenapine = 190; N placebo = 189) | 6 | 14
  Days 15 - 21 (N asenapine = 184; N placebo = 175) | 3 | 10
  Days 22 - 28 (N asenapine = 181; N placebo = 165) | 5 | 11
  Days 29 - 35 (N asenapine = 176; N placebo = 154) | 0 | 11
  Days 36 - 42 (N asenapine = 176; N placebo = 143) | 3 | 7
  Days 43 - 49 (N asenapine = 173; N placebo = 136) | 7 | 7
  Days 50 - 56 (N asenapine = 166; N placebo = 129) | 0 | 3
  Days 57 - 63 (N asenapine = 166; N placebo = 126) | 3 | 4
  Days 64 - 70 (N asenapine = 163; N placebo = 122) | 1 | 2
  Days 71 - 77 (N asenapine = 162; N placebo = 120) | 0 | 4
  Days 78 - 84 (N asenapine = 162; N placebo = 116) | 4 | 3
  Days 85 - 91 (N asenapine = 158; N placebo = 113) | 5 | 8
  Days 92 - 98 (N asenapine = 153; N placebo = 105) | 2 | 4
  Days 99 - 105 (N asenapine = 150; N placebo = 100) | 0 | 2
  Days 106 - 112 (N asenapine = 150; N placebo = 98) | 1 | 1
  Days 113 - 119 (N asenapine = 149; N placebo = 97) | 1 | 8
  Days 120 - 126 (N asenapine = 148; N placebo = 88) | 0 | 1
  Days 127 - 133 (N asenapine = 148; N placebo = 87) | 2 | 0
  Days 134 - 140 (N asenapine = 146; N placebo = 86) | 0 | 1
  Days 141 - 147 (N asenapine = 145; N placebo = 84) | 3 | 1
  Days 148 - 154 (N asenapine = 142; N placebo = 82) | 1 | 3
  Days 155 - 161 (N asenapine = 141; N placebo = 78) | 1 | 3
  Days 162 - 168 (N asenapine = 139; N placebo = 75) | 2 | 1
  Days 169 - 175 (N asenapine = 137; N placebo = 73) | 2 | 1
  Days 176 - 182 (N asenapine = 135; N placebo = 71) | 0 | 1
  Days 183 - 189 (N asenapine = 75; N placebo = 39) | 0 | 0
  Days 190 - 196 (N asenapine = 9; N placebo = 9) | 0 | 0
  Days 197 - 203 (N asenapine = 2; N placebo = 2) | 0 | 0
  Days 204 - 210 (N asenapine = 0; N placebo = 1) | 0 | 0

ADVERSE EVENTS:
Time Frame: Prior to randomization to the double-blind period, there was a 26 week open-label phase where 700 subjects received at least one dose of open-label asenapine (out of 831 initially enrolled).
Description: During the first 4 weeks of the open-label period, subjects could cross titrate. The target dose of asenapine was 10 mg twice daily by week 1. Only subjects who had continued stable presentation of symptoms during open-label phase were randomized into the double-blind phase (into Asenapine or Placebo arm). Remainder of subjects were not randomized.
Groups:
- Asenapine: Adverse Events for the Double Blind Period. Subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1), followed by asenapine 5 or 10 mg sublingual twice daily for 26 weeks in the double blind phase.
- Placebo: Adverse Events for the Double Blind Period. Subjects received 26 weeks of open label asenapine treatment (cross titration period up to first 4 weeks, with target dose of 10 mg twice daily by week 1), followed by matching placebo sublingual twice daily for 26 weeks during the double-blind phase.
- Asenapine During Open-Label Phase and Not Randomized: Adverse Events for the Open-Label period. The 'Asenapine During Open-Label Phase & Not Randomized' Group includes subjects who received >= 1 dose of asenapine during the 26 week open-label phase, and did NOT continue to double-blind phase.
Arm/Group | Asenapine | Placebo | Asenapine During Open-Label Phase and Not Randomized
Serious Adverse Events (participants affected / at risk) | 6/194 | 22/192 | 39/314
Other Adverse Events (participants affected / at risk) | 121/194 | 127/192 | 170/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=194) | Placebo (N=192) | Asenapine During Open-Label Phase and Not Randomized (N=314)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOTHERMIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
ADNEXITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
EXTERNAL EAR CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPINAL CORD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BLOOD GLUCOSE DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
POOR QUALITY SLEEP (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
TARDIVE DYSKINESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
HALLUCINATION, VISUAL (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
HOMICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
PARANOIA (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
SCHIZOPHRENIA (Psychiatric disorders) | 2 (2) | 9 (9) | 10 (11)
SCHIZOPHRENIA, PARANOID TYPE (Psychiatric disorders) | 2 (2) | 7 (7) | 11 (11)
SCHIZOPHRENIA, UNDIFFERENTIATED TYPE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
THINKING ABNORMAL (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
BALANOPOSTHITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asenapine (N=194) | Placebo (N=192) | Asenapine During Open-Label Phase and Not Randomized (N=314)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 4 (5) | 10 (11) | 11 (11)
NAUSEA (Gastrointestinal disorders) | 9 (10) | 10 (10) | 15 (15)
WEIGHT DECREASED (Investigations) | 13 (13) | 21 (24) | 3 (3)
WEIGHT INCREASED (Investigations) | 28 (30) | 21 (23) | 11 (11)
AKATHISIA (Nervous system disorders) | 13 (23) | 13 (20) | 21 (32)
HEADACHE (Nervous system disorders) | 21 (33) | 19 (28) | 19 (45)
PARKINSONISM (Nervous system disorders) | 10 (14) | 12 (18) | 12 (19)
SEDATION (Nervous system disorders) | 10 (14) | 10 (13) | 12 (16)
SOMNOLENCE (Nervous system disorders) | 31 (43) | 33 (47) | 54 (65)
AGITATION (Psychiatric disorders) | 12 (13) | 19 (20) | 24 (29)
ANXIETY (Psychiatric disorders) | 25 (32) | 27 (46) | 34 (48)
DELUSION (Psychiatric disorders) | 2 (2) | 12 (15) | 12 (13)
DEPRESSION (Psychiatric disorders) | 13 (14) | 9 (12) | 15 (20)
HALLUCINATION (Psychiatric disorders) | 2 (2) | 13 (15) | 6 (6)
INSOMNIA (Psychiatric disorders) | 39 (48) | 47 (64) | 42 (56)
SCHIZOPHRENIA (Psychiatric disorders) | 8 (8) | 25 (32) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will be provided an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed.

Materials for intended disclosure must be provided to sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, then the disclosure must be delayed for a period not to exceed an additional 60 days.